CLINICAL TRIAL: NCT06737887
Title: The Effect of Preoperative Stoma Simulation on Anxiety and Postoperative Adaptation: A Randomised Controlled Trial
Brief Title: The Effect of Preoperative Stoma Simulation on Anxiety and Postoperative Adaptation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hatice Merve Alptekin, Research Assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/410
Record Dates: First submitted 2024-12-11; First posted 2024-12-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-03

CONDITIONS: Colostomy - Stoma; Ileostomy - Stoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stoma simulation group (Experimental): 1. Patients are informed about the study 24 hours before surgery.
  2. The patient is given a "patient information form" and "The State-Trait Anxiety Inventory".
  3. The stoma simulation is started.
  4. The stoma simulation is ended on the morning of the surgery and the patient's state anxiety is measured.
  5. During the discharge, the patient's adaptation to the stoma is evaluated using the Ostomy Adjustment Inventory.
  6. 1 months after surgery, the patient's adaptation to the stoma is evaluated again using the Ostomy Adjustment Inventory.
  Interventions: Other: Stoma simulation
- Control group (No Intervention): 1. Patients are informed about the study 24 hours before the surgery.
  2. The patient is given a "patient information form" and "The State-Trait Anxiety Inventory".
  3. The patient's state anxiety is measured on the morning of the surgery.
  4. During the discharge, the patient's adaptation to the stoma is evaluated using the Ostomy Adjustment Inventory.
  5. 3 months after the surgery, the patient's adaptation to the stoma is evaluated again using the Ostomy Adjustment Inventory.

INTERVENTIONS:
Other: Stoma simulation — Patients who will undergo stoma surgery will have an intervention one day before the surgery. The adapter will be cut to an estimated stoma size, heated by rubbing with hands and adapted to the skin by applying stoma paste. The patient will be asked to place their hand on the adapter and apply pressure. Then, the stoma bag filled with tissues and water and the adapter will be combined. The patient will be informed that they should not hesitate to do any activity that they will spend 24 hours with the stoma bag. The patient will be provided with the opportunity to go to the toilet, eat, sleep and experience all their daily activities with the stoma. It allows patients to experience the stoma bag by putting it on 24 hours before the surgery. In this way, patients know that they will not encounter any surprises after the surgery.
  Arms: Stoma simulation group

SUMMARY:
The majority of patients (60-70%) develop high levels of anxiety before surgery. Surgical patients may experience feelings of anxiety due to insufficient information and counseling before surgery and potential changes in the body caused by surgery. Fears include (but are not limited to) not waking up from anesthesia, not being able to return to previous work and family life, and adaptation concerns regarding new processes after surgery. Patients with fear of complications experience preoperative anxiety four times more than other patients. Other factors affecting preoperative anxiety were determined to be waiting for a long time before surgery, not knowing what will happen during surgery, losing control of the body, not receiving sufficient social support, being exposed to medical errors, and encountering undesirable health outcomes after surgery. The changes that will occur in the body and lifestyle after stoma surgery scare patients and cause them to feel anxiety in the pre-operative period. Despite significant developments in stoma care products and the increase in the number of nurses specialized in stoma care in recent years, the majority of patients experience problems with compliance. For this reason, the compliance of stoma patients with stoma life is increasingly the subject of clinical trials and epidemiological studies. In our country, studies conducted to determine the problems experienced by stoma individuals regarding compliance with stoma and social life are limited. Nursing interventions are recommended to reduce patients' anxiety and increase their compliance with stoma after surgery. This study aims to evaluate the effect of stoma simulation performed preoperative surgery on the patient's anxiety level and postoperative stoma compliance.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are planned for elective stoma surgery,
* Are between the ages of 18-65,
* Can speak Turkish,
* Can read and write,
* Are conscious,
* Are willing to participate in the study will be included.

Exclusion Criteria:

* Patients with speech or hearing impairments,
* Those who have had urostomy surgery,
* Those who have a psychological diagnosis or are taking medication,
* Those who need intensive care after surgery,
* Those whose stoma was closed during the study,
* Those who have complications in the peristomal area,
* Patients who have had stoma surgery before will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2027-01-02 (Estimated); Primary Completion 2027-02-02 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 24 hours before surgery and 30 minutes before surgery
  The State-Trait Anxiety Inventory consists of two separate dimensions: state anxiety (STAI-I) and trait anxiety (STAI-II), and these dimensions aim to measure individuals' anxiety states in different contexts. The scale consists of 40 items in total; 20 items measure state anxiety and the other 20 items measure trait anxiety. Both scales are scored between 20-80, and as the score increases, the level of anxiety increases. The State-Trait Anxiety Inventory is administered 24 hours before surgery. The patient's state anxiety is measured 30 minutes before surgery.

SECONDARY OUTCOMES:
Stoma adaptation | the morning of the patient's discharge (7th day of surgery) and 1 months after surgery
  The patient's adaptation to the stoma is assessed with the Ostomy Adjustment Inventory. The scale consists of 23 items and four sub-dimensions. The sub-dimensions are acceptance, anger, anxiety/worry, and social adaptation. The lowest score on the scale is 0, and the highest is 92. A high score on the scale indicates that the individual's adaptation to the stoma is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Istanbul Medical Faculty Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No